CLINICAL TRIAL: NCT06653621
Title: Effect of Bupivacaine Liposomes or Bupivacaine for Femoral Triangle or Adductor Block on Analgesia After Total Knee Replacement: a Prospective, Single-center, Simple Randomized, Active-controlled, Single-blind, 2x2 Factorial Design Clinical Study
Brief Title: Effect of Bupivacaine Liposomes or Bupivacaine for Femoral Triangle or Adductor Block on Analgesia After Total Knee Replacement
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wei Mei, clinical professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: TJ-IRB202409095
Record Dates: First submitted 2024-10-15; First posted 2024-10-22 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Knee Arthropathy; Knee Arthritis
Keywords: Knee Arthropathy; liposome bupivacaine; femoral nerve block; adductor canal block
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: This study utilizes a factorial interventional design, where participants undergoing total knee arthroplasty surgery will be allocated into four separate groups. Group one will receive liposomal bupivacaine plus bupivacaine as a regional anesthetic for adductor block, the group two will receive bupivacaine for adductor block; the group three will receive liposomal bupivacaine plus bupivacaine as a regional anesthetic for femoral nerve block ; Group four will receive bupivacaine as a regional anesthetic for femoral nerve block .Two types of interventions are involved, namely, choice of anesthesia mode (2 levels: adductor block, femoral triangle block) and anesthetic administration (2 levels: bupivacaine liposomes and bupivacaine mixture, bupivacaine).The study aims to compare the analgesic efficacy, duration of pain relief, opioid consumption, between the four groups .
Who Masked: Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor) . Given the distinct visual appearance of the liposomal bupivacaine (milky white) and bupivacaine (transparent), a double-blind study design is not feasible. Consequently, this study employs a single-blind approach where neither participants nor outcome assessors will be aware of treatment allocation. Healthcare providers administering the study drug will be aware of the treatment group assignment. Rigorous procedures will be implemented to minimize potential bias, including standardized outcome assessment tools, blinded data entry, and independent data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- adductor block+ Bupivacaine liposomes and bupivacaine mixture (Experimental): The patient underwent ultrasound-guided bupivacaine liposome mixture single adductor block during anesthesia induction room for analgesia after total knee arthroplasty .
  Interventions: Drug: Bupivacaine liposome; Procedure: Nerve block mode : adductor block
- adductor block+ bupivacaine (Active Comparator): The patient underwent ultrasound-guided bupivacaine single adductor block during anesthesia induction room for analgesia after total knee arthroplasty
  Interventions: Procedure: Nerve block mode : adductor block; Drug: Bupivacaine
- femoral triangle block + Bupivacaine liposomes and bupivacaine mixture (Experimental): The patient underwent ultrasound-guided bupivacaine liposome mixture single femoral triangle block during anesthesia induction room for analgesia after total knee arthroplasty .
  Interventions: Drug: Bupivacaine liposome; Procedure: Nerve block mode: femoral triangle block
- femoral triangle block + bupivacaine (Active Comparator): The patient underwent ultrasound-guided bupivacaine single femoral triangle block during anesthesia induction room for analgesia after total knee arthroplasty .
  Interventions: Drug: Bupivacaine; Procedure: Nerve block mode: femoral triangle block

INTERVENTIONS:
Drug: Bupivacaine liposome — Subjects receive liposomal bupivacaine as a regional anesthetic for femoral triangle block or adductor block under ultrasound guidance.
  Other Names: L
  Arms: adductor block+ Bupivacaine liposomes and bupivacaine mixture; femoral triangle block + Bupivacaine liposomes and bupivacaine mixture
Procedure: Nerve block mode : adductor block — Subjects receive liposomal bupivacaine or bupivacaine as a regional anesthetic for adductor block under ultrasound guidance.
  Other Names: A
  Arms: adductor block+ Bupivacaine liposomes and bupivacaine mixture; adductor block+ bupivacaine
Drug: Bupivacaine — Subjects receive bupivacaine as a regional anesthetic for femoral triangle block or adductor block under ultrasound guidance.
  Other Names: B
  Arms: adductor block+ bupivacaine; femoral triangle block + bupivacaine
Procedure: Nerve block mode: femoral triangle block — Subjects receive liposomal bupivacaine or bupivacaine as a regional anesthetic for femoral triangle block under ultrasound guidance.
  Other Names: F
  Arms: femoral triangle block + Bupivacaine liposomes and bupivacaine mixture; femoral triangle block + bupivacaine

SUMMARY:
The purpose of this study was to investigate the effect of bupivacaine liposomes on postoperative pain in TKA ( total knee replacement ) patients.The main questions answered are:

1. Is bupivacaine liposomes superior to bupivacaine in femoral triangle block or adductor block in terms of 72 hours opioid consumption after knee replacement
2. Which block method(Femoral triangle block or adductor block) combined with bupivacaine liposome was more effective in alleviating pain score and 72 hours opioid consumption after total knee surgery.

investigators will investigate the effect of bupivacaine liposomes combined with bupivacaine and pure bupivacaine on pain after total knee arthroplasty using femoral triangle block or adductor block.

Participants will:

1. Receive liposomal bupivacaine or bupivacaine as a regional anesthetic for femoral triangle block or adductor block under ultrasound guidance.
2. Undergo total knee replacement surgery under spinal anesthesia.
3. Follow-up within 72 hours after surgery , opioid consumption, NRS score, PCA（Patient controlled analgesia，PCA） data, first postoperative remedial analgesia time, quadriceps muscle strength and complications were recorded

DETAILED DESCRIPTION:
The patients received femoral triangle block plus iPACK(infiltration between popliteal artery and capsule of knee) block or adductor canal block plus iPACK block during induction .

The local anesthetic formulation was bupivacaine (0.75% bupivacaine hydrochloride 10ml+ normal saline 20ml) or bupivacaine liposome (0.75% bupivacaine hydrochloride 10ml+ bupivacaine liposome 20ml(266mg)).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ASAI-ⅲ
2. Receive a unilateral initial TKA
3. Age 18-80 years old -

Exclusion Criteria:

1. Bilateral TKA surgery
2. TKA revision surgery
3. Contraindications for nerve block and intraspinal anesthesia
4. Allergies to local anesthetics
5. Diabetic neuropathy
6. Patients who are unable to cooperate with the evaluation
7. Chronic use of opioid analgesics
8. BMI≥35kg/cm2
9. Cases of lumbar anesthesia failure requiring general anesthesia surgery
10. Cases of nerve block failure

    -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-11-05 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption 72 hours after surgery | this outcome will be monitored and recorded within 72 hours postoperatively
  This primary outcome entails tracking and assessing the total opioid consumption by participants following total knee replacement surgery. The evaluation includes quantifying the amount of opioids prescribed and consumed by participants for pain management post-surgery. Opioid medications administered will be converted to morphine equivalents based on established conversion ratios. By analyzing overall opioid consumption, the study aims to evaluate the efficacy of the interventions in managing postoperative pain.

SECONDARY OUTCOMES:
Pain intensity | Pain intensity will be measured at 8 time points: 6 hours, 12 hours, 18 hours and 24 hours 36 hours, 48 hours, 60 hours, 72 hours post-surgery
  Pain intensity will be assessed using the Numerical Rating Scale (NRS), a 0-10 scale where 0 represents no pain and 10 represents the worst imaginable pain
Time to First Rescue Analgesic | 72 hours after surgery
  Time to first rescue analgesic will be recorded as the interval from the end of the surgery to the administration of the first dose of rescue analgesic medication postoperatively.
Total opioid dosage and PCA times | Total opioid dosage and PCA times were recorded at 8 time points: 6 hours, 12 hours, 18 hours and 24 hours 36 hours, 48 hours, 60 hours, 72 hours post-surgery
  The evaluation includes quantifying the amount of opioids prescribed and consumed PCA times by participants for pain management post-surgery.
Quadriceps muscle strength | 24.48,72 hours after surgery
  The quadriceps muscle strength is measured with a hand-held dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: wei mei, MD, Principal Investigator — Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Lingli DENG, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chuan A, Lansdown A, Brick KL, Bourgeois AJG, Pencheva LB, Hue B, Goddard S, Lennon MJ, Walters A, Auyong D; Continuous Catheters in Adductor Canal versus Femoral Triangle (The CAFE study) investigators. Adductor canal versus femoral triangle anatomical locations for continuous catheter analgesia after total knee arthroplasty: a multicentre randomised controlled study. Br J Anaesth. 2019 Sep;123(3):360-367. doi: 10.1016/j.bja.2019.03.021. Epub 2019 May 2. PMID 31056239
- [Background] Song L, Li Y, Xu Z, Geng ZY, Wang DX. Comparison of the ultrasound-guided single-injection femoral triangle block versus adductor canal block for analgesia following total knee arthroplasty: a randomized, double-blind trial. J Anesth. 2020 Oct;34(5):702-711. doi: 10.1007/s00540-020-02813-8. Epub 2020 Jun 12. PMID 32533332